CLINICAL TRIAL: NCT02487420
Title: Trapsgewijze Ei-tolerantie-inductie Bij Kippenei-allergische Kinderen (TETI Studie)
Brief Title: Gradual Egg-tolerance Induction in Hen's Egg Allergic Children
Acronym: TETI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dominque Bullens (Other)
Collaborators: Jessa Hospital (Other); Algemeen Ziekenhuis Maria Middelares (Other); Imelda Hospital, Bonheiden (Other); AZ Sint-Jan AV (Other)
Responsible Party: Sponsor-Investigator, Dominque Bullens, MD, PhD, Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: S57588
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Egg Hypersensitivity
MeSH Terms: conditions — Egg Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 18m (Other): arm 18m: 6 months between step 1 and step 2; 6 months between step 2 and step 3, 3 months between all other steps step by step gradual introduction of egg containing food products during 18 months, unless next step can not be taken
  Interventions: Behavioral: shorter or longer period of specific dietary restrictions
- arm 30 m (Other): arm 30m: 9 months between step 1 and step 2; 9 months between step 2 and step 3, 6 months between all other steps step by step gradual introduction of egg containing food products during 30 months, unless next step can not be taken
  Interventions: Behavioral: shorter or longer period of specific dietary restrictions

INTERVENTIONS:
Behavioral: shorter or longer period of specific dietary restrictions — step by step gradual introduction of egg containing food products

SUMMARY:
1. The investigators here want to test the hypothesis that a total period of 18 months of gradual open introduction of a certain egg product with regard to full egg tolerance induction is not inferior when compared to a total period of 30 months gradual open introduction of a certain egg product (see steps for the specific egg products) after tolerance for baked egg has been obtained.
2. The investigators also want to define step-specific 'tolerance-failures' and study the relevance of specific IgE to specific egg components to predict failures at each step.

DETAILED DESCRIPTION:
1. The investigators here want to test the hypothesis that a total period of 18 months of gradual open introduction of a certain egg product with regard to full egg tolerance induction is not inferior when compared to a total period of 30 months gradual open introduction of a certain egg product (see steps for the specific egg products) after tolerance to baked egg has been obtained.
2. The investigators also want to define step-specific 'tolerance-failures' and study the relevance of specific IgE to specific egg components to predict failures at each step.

Step 1: open baked egg test passed (either at home or in the hospital): this is routine clinical practice; afterwards daily intake of increasing amounts of heated egg (amounts to be noted in diary)

Step 2: open provocation test at home with hard-boiled egg, both hen's egg white and yolk, passed; afterwards weekly intake of either hard-boiled egg white or yolk or both (amounts and days to be noted in diary)

Step 3: open provocation test at home with waffles, omelet, pan cake or scrambled egg passed; afterwards weekly or two-weekly intake of one of these specific preparation forms or of the previous preparation forms (amounts, days and preparation to be noted in diary)

Step 4: open provocation test at home with fried or poached egg or softly boiled egg with liquid yolk; afterwards regular intake of one of these preparation forms or one of the prior steps (amounts, days and preparation to be noted in diary)

Step 5: open provocation test at home with raw egg: eg. In chocolate mousse; mayonnaise or tiramisu; afterwards unlimited intake of all egg containing preparation forms (for 3 months in both groups to be noted in the diary)

If tolerance to a certain step is not yet present (this is: if any reaction occurred during the months registered between two steps), the next step will be postponed. The number of failures (any reaction in relation to egg ingestion), the type of reaction and the additional time period necessary before the next step can be taken, will be recorded. After each time period, the investigators will measure specific IgE to hen's egg white and to Gal d 1, as standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Children (1-18y) had or have a clinical diagnosis of IgE mediated hen's egg allergy based on positive history as well as skin prick testing and/or specific IgE detection by CAPtest in an allergy clinic
2. Children are at least 12 months old before introduction of heated egg is considered
3. Children did not suffer from a moderate-to-severe anaphylaxis due to egg-ingestion at presentation
4. Children have specific IgE levels to Gal d 1 below 1.2 kU/mL or passed cake provocation test -

Exclusion Criteria:

1. Children had a moderate-to severe anaphylaxis due to egg ingestion
2. Children are younger than 12 months old at the moment of passing heated egg open provocation test
3. Parents are not able or not willing to test a certain step in the tolerance induction at home -

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
time to complete egg tolerance | 18 to 30 months
  raw egg tolerance (eg in chocolate mousse)

SECONDARY OUTCOMES:
Measurement of specific IgE to egg white components to predict complete egg tolerance | 18 to 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Dominique MA Bullens, MD, PhD, Principal Investigator — UZ Leuven
Locations (6):
- Belgium (6):
  - University Hospital of Leuven, Leuven, Vlaams-Brabant
  - Imelda Hospital, Bonheiden, Bonheiden
  - Sint-Jan, Bruges
  - Algemeen Ziekenhuis Maria Middelares, Ghent
  - Jessa Hospital, Hasselt
  - Sint-Jan, Ostend

IPD SHARING:
Plan to Share IPD: No
data will be analysed and grouped before release